CLINICAL TRIAL: NCT04873518
Title: 3D-Transition Study: Challenges and Resources of Children and Their Families During the Transition From Preschool to School, in a Pregnancy Cohort
Brief Title: 3D-Transition: Challenges and Resources of Children and Their Families During the Transition From Preschool to School
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Université de Sherbrooke (Other); CHU de Quebec-Universite Laval (Other); Université de Montréal (Other); Laval University (Other)
Responsible Party: Principal Investigator, Jean Séguin, Researcher, St. Justine's Hospital
Other Study IDs: MP-21-2017-1461; PJT-148551 (Other Grant/Funding Number: Canadian Institutes for Health Research); PJT-165824 (Other Grant/Funding Number: Canadian Institutes for Health Research); CRI-88413 (Other Grant/Funding Number: Canadian Institutes for Health Research)
Record Dates: First submitted 2021-04-13; First posted 2021-05-05 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Issue; Externalizing Behavior Problems; Internalizing Behavior Problems; Cognitive Development; Neurodevelopmental Disorders; Academic Achievement
Keywords: longitudinal; cohort-sequential
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary hormones in a subsample of 382 children
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: These are the eldest children who entered kindergarten in September 2016.
- Cohort 2: These children entered kindergarten in September 2017.
- Cohort 3: These are the youngest children who entered kindergarten in September 2018

SUMMARY:
The 3D-Transition study is a follow-up of the 3D Cohort pregnancy study (NCT03113331, which covered from the 1st trimester of pregnancy to age 2 years) as the children transition into kindergarten and first grade. It aims at clarifying prenatal and preschool predictors of challenging and successful transitions to school as measured by mental health and academic outcomes.

DETAILED DESCRIPTION:
Broad goal: This study seeks to understand how early vulnerabilities (externalizing or internalizing symptoms, or low neurodevelopmental/academic skills) turn into a rate of 10-15% of externalizing and internalizing mental health problems in school-aged children.

Rationale: Several lines of research guide this study. Functional impairments emerge for some children challenged by the transition to kindergarten and grade school. This risk is also thought to be programmed very early in life through cumulative early perinatal and psychosocial adversity. Further, interactions between the child, family and school environment during the transition may mitigate future impairments and this may be different for boys and girls. Finally, stress regulation mechanisms during the transition seem linked to early child vulnerabilities. This design allows us to contrast any combination of these mechanisms.

Aims: This study will clarify the role of:

1. a mismatch between some child preschool vulnerability (externalizing, or internalizing symptoms, or low neurodevelopmental/academic skills) and the challenges of the transition from preschool to formal schooling;
2. the experience of perinatal adversity and home chaos during child first years;
3. supportive environments (high quality families or schools) during the school transition, and child sex; and
4. the child stress response to the school transition, as assessed through salivary cortisol.

Method: Building on an existing pregnancy cohort (NCT03113331, which was structured around a triadic (mother-partner-child) framework, and which covered from the 1st trimester of pregnancy to age 2 years), the investigators have followed at least once 939 of 1551 families that agreed to a further follow-up past the initial study. Children in this cohort, who were seen in 3 waves based on age on September 30th, entered kindergarten in the fall of 2016, 2017, and 2018, respectively. A cohort-sequential longitudinal research design spanning pre-kindergarten to 2nd grade (ages 4 to 8 years), was implemented to follow each wave 6 times over 4 years. Cascade models will be used to address aims 1-3. The stress hormone cortisol will be examined on 11 days spread over a 16 months period for a subsample of 384 children to address aim 4, using growth curves models. This design is well suited and sufficiently powered to examine change processes over time, controlling for potential differences in waves and time of measurement effects.

Additional data: The Research Ethics Committee authorized two Corona Virus (COVID-19) supplemental data collections without additional consent for the spring of 2020 and the spring of 2021. However, cohorts 1 and 2, which had completed participation in 2019 and 2020, were re-consented, and this extended the maximum age range to 10 and 9 years, respectively. As of 2022-05-03 investigators are in the process of requesting approval for an additional COVID-19 follow-up.

Expected outcomes: Public health interventions are being put in place to help children manage the transition to school on the basis of little evidence. This longitudinal research will provide a greater understanding of individual and environmental factors linked to children's adaptation during the perinatal period and transitions to school. As such, mental health prevention research will be better informed on the developmental timing of individual and environmental targets that need to be considered in a developmental framework.

ELIGIBILITY:
Inclusion Criteria:

* All participating families from Clinical Trials NCT03113331 who had accepted a follow-up past the original pregnancy to age 2-years time span of that protocol.

Exclusion Criteria:

* None for this follow up. See Clinical Trials NCT03113331 for original exclusion criteria.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: General population sample from the main university hospitals affiliated with the province of Québec, Canada's 4 faculties of medicine between November 2010 and March 2013, included.
Sampling Method: Non-Probability Sample
Enrollment: 939 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-12-21 (Estimated); Study Completion 2022-12-21 (Estimated)

PRIMARY OUTCOMES:
Mental health: Change in child mental health represented by one latent symptom score of the overarching category: externalizing symptoms. | Six times across 4 years, in the spring during Pre-Kindergarten, then in the fall and spring of Kindergarten and Grade 1, then in the spring of Grade 2
  The latent factor will be based on three informants which provide these mental health symptom ratings: mother-, father-, and teacher-reports as measured with age-appropriate non-overlapping items from the externalizing symptoms scales of:
  i) the Strengths and Difficulties Questionnaire (SDQ) ii) the Child Behavior Checklist (CBCL) iii) the Behavior scale of the Quebec Longitudinal Study of Child Development (QLSCD).
Mental health: Change in child mental health represented by one latent symptom score of the overarching category: internalizing symptoms. | Six times across 4 years, in the spring during Pre-Kindergarten, then in the fall and spring of Kindergarten and Grade 1, then in the spring of Grade 2
  The latent factor will be based on three informants which provide these mental health symptom ratings: mother-, father-, and teacher-reports as measured with age-appropriate non-overlapping items from the externalizing symptoms scales of:
  i) the Strengths and Difficulties Questionnaire (SDQ) ii) the Child Behavior Checklist (CBCL) iii) the Behavior scale of the Quebec Longitudinal Study of Child Development (QLSCD).
Neurodevelopment - Change in executive function | Yearly, across 3 years: in Pre-Kindergarten, Kindergarten and Grade 1
  Change in one latent factor score of executive function based on the following tasks:
  1. Dimensional Change Card Sort (DCCS) measuring degree of cognitive flexibility
  2. Random Object Span Task (ROST), a child version of the Self-Ordered Pointing (SOP) test measuring degree of working memory.
  3. Wechsler's Digit Span subtest measuring degree of working memory.
Neurodevelopment - Change in visuo-spatial ability | Yearly, across 3 years: in Pre-Kindergarten, Kindergarten and Grade 1
  Change in visuo-spatial ability based on the Wechsler's Block Design subtest.
Neurodevelopment - Change in visuo-motor integration | Yearly, across 2 years: in Pre-Kindergarten and in Kindergarten
  Change on the Beery Visuo-Motor integration subtest.
Neurodevelopment - Change in social cognition | Yearly, across 3 years: in Pre-Kindergarten, Kindergarten and Grade 1
  Change in social cognition based on a latent factor of 1st and 2nd order Theory Of Mind (TOM) tests.
Neurodevelopment - Change in emotional development | Yearly, across 3 years: in Pre-Kindergarten, Kindergarten and Grade 1
  Change on the Pons and Harris (2000) Test of Emotion Comprehension (TEC) score.
Academic skills scores - Change in school readiness | Yearly, across 2 years: in Pre-Kindergarten and Kindergarten
  Change in the total score of The Lollipop Test comprising 4 dimensions: 1) Identification of Colors and Shapes, and Copying Shapes, 2) Picture Description, Position, and Spatial Recognition, 3) Identification of Numbers, and Counting, and 4) Identification of Letters, and Writing.
Academic skills scores- Change in Number Knowledge abilities | Yearly, across 3 years: in Pre-Kindergarten, Kindergarten and Grade 1
  Change in a score combining The Number Knowledge Test (NKT) and the Mathematics subtest of the Canadian Achievement Test (CAT).
Academic skills scores - Change in receptive vocabulary | Yearly, across 3 years: in Pre-Kindergarten, Kindergarten and Grade 1
  Change in the total score of the Peabody Picture Vocabulary Test (PPVT) in French or English versions.
Academic skills scores - Change in Reading ability | Grade 1 only
  The Kaufman Assessment Battery for Children (K-ABC) reading ability test score in French or English versions.
Academic skills scores - Change in academic performance. | Yearly, across 2 years: in Grades 1 and 2
  Change in teacher reports on child academic achievement.
Change in Morning and evening salivary cortisol levels | Pre-Kindergarten to Grade 1 (Across a 16 months period from June in Year 1 to September in Year 2)
  A subsample of 382 (out of 400 targeted) from cohorts 2 and 3 participated in a measurement burst design of 11 measurement days (2 samples/day), in June and August preceding entry into kindergarten (baseline), then twice one week apart at kindergarten entry in early September, then first Wednesday in each of November, February, and April. The following June, August, and early September measures were then repeated as the children moved towards entry to 1st grade.

CONTACTS AND LOCATIONS:
Overall Officials: Jean R. Séguin, Ph.D., Principal Investigator — CHU Ste-Justine Research Center and Université de Montréal; Sophie Parent, Ph.D., Principal Investigator — CHU Ste-Justine Research Center and Université de Montréal; Natalie Castellanos-Ryan, Ph.D., Principal Investigator — CHU Ste-Justine Research Center and Université de Montréal
Locations (3):
- Canada (3):
  - CHU Ste-Justine Research Center, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The procedures by which de-identified data will be accessible are being clarified as rules and regulations are currently under study in this jurisdiction. In the meantime the investigators can be contacted for updates - see "More information"
Time Frame: Partial data from earlier waves may be available upon request. The bulk of the data should be available by March 2023.
Access Criteria: Data are under the jurisdiction of the Centre Hospitalier Universitaire (CHU) Ste-Justine Research Ethics Committee and subject to current provincial and national privacy laws guiding their ethical use in Québec, Canada. To submit a request, please visit the 3D-Cohort Study website or contact the principal investigator.
URL: http://www.irnpqeo.ca/en/researchers/

REFERENCES:
- [Background] Parent S, Lupien S, Herba CM, Dupere V, Gunnar MR, Seguin JR. Children's cortisol response to the transition from preschool to formal schooling: A review. Psychoneuroendocrinology. 2019 Jan;99:196-205. doi: 10.1016/j.psyneuen.2018.09.013. Epub 2018 Sep 14. PMID 30253327
- [Background] Rioux C, Parent S, Castellanos-Ryan N, Archambault I, Boivin M, Herba CM, Lupien SJ, Marc I, Muckle G, Fraser WD, Seguin JR. The 3D-Transition Study: Objectives, Methods, and Implementation of an Innovative Planned Missing-Data Design. Am J Epidemiol. 2021 Nov 2;190(11):2262-2274. doi: 10.1093/aje/kwab141. PMID 33987638
- [Result] Leblond M, Parent S, Castellanos-Ryan N, Lupien SJ, Fraser WD, Seguin JR. Transition from preschool to school: Children's pattern of change in morning cortisol concentrations. Psychoneuroendocrinology. 2022 Jun;140:105724. doi: 10.1016/j.psyneuen.2022.105724. Epub 2022 Mar 14. PMID 35325645